CLINICAL TRIAL: NCT01399320
Title: Ghnnam Excision Technique for Pilonidal Sinus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Wagih Mommtaz Ghnnam, Mansoura faculty of medicine general surgery department
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MansouraU
Record Dates: First submitted 2011-07-19; First posted 2011-07-21 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2008-08

CONDITIONS: Pilonidal Sinus; Surgical Wound; Dressing by Cyanoacrylate
Keywords: Pilonidal disease; Excision; cyanoacrylate
MeSH Terms: conditions — Pilonidal Sinus; Surgical Wound | interventions — Cyanoacrylates; Enbucrilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cyanoacrylate dressing,excesion (Experimental): we excise the sinus tip then apply cyanoacrylate dressing and watch for healing
  Interventions: Procedure: cyanoacrylate

INTERVENTIONS:
Procedure: cyanoacrylate — excision of the sinus under local anesthesia the packing of the wound by cyanoacrylate dressing
  Other Names: histoacryl

SUMMARY:
Pilonidal disease is a common disorder of the sacrococcygeal region. It comprises a variety of problems, including infection/abscess and the development of a chronic sinus cavity.here we try a minimmally invasive method for managing such condition

DETAILED DESCRIPTION:
Pilonidal disease is a common disorder of the sacrococcygeal region. It comprises a variety of problems, including infection/abscess and the development of a chronic sinus cavity. Incidence varies across countries and races .The cause remains controversial. Both congenital and acquired causes have been postulated Excision with a simple lay-open or performing marsupialization both result in a midline wound that takes several weeks to heal and there is a significant recurrence rate because of the open portal for hair insertion.so here we apply a new minimally invasive excision with cyanoacrylate dressing

ELIGIBILITY:
Inclusion Criteria:

* any patient with pilonidal sinus

Exclusion Criteria:

* pilonidal abscess or sever acute inflammation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-08; Primary Completion 2009-09 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
healing of the sinus | 1 month

SECONDARY OUTCOMES:
recurrence | 1 year
  no recurrence
wound infection | 3-6 months
  occurrence of wound sepsis
patient satisfaction | 3 months
  patient satisfied with the procedure

CONTACTS AND LOCATIONS:
Overall Officials: wagih m ghnnam, MD, Principal Investigator — mansoura faculty of medicine general surgery department
Locations (1):
- Mansoura Faculty of Medicine, Al Mansurah, Dakahlia Governorate, Egypt